CLINICAL TRIAL: NCT06648356
Title: Short Term Effects of Proprioceptive Neuromuscular Facilitation Combined With Neuromuscular Electrical Stimulation in Young Basketball Players: a Randomized Clinical Trial.
Brief Title: Effects of Combining PNF With NMES in Young Basketball Players
Acronym: PNF+NMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Professor, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIVERSITY CARDENAL HERRERA-86
Record Dates: First submitted 2024-10-14; First posted 2024-10-18 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Hamstring Flexibility
Keywords: hamstring flexibility; vertical jump; basketball; Propioceptive Neuromuscular Facilitation; Neuromuscular Electrical Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- contract-relax proprioceptive neuromuscular facilitation (crPNF) (Active Comparator): Participants in this group performed a stretching protocol using contract-relax proprioceptive neuromuscular facilitation (crPNF). The participants are placed in a long sitting position with maximum knee extension possible until a moderate-strong stretch sensation is felt, without pain. The stretch lasts for 20 seconds, followed by a maximal voluntary isometric contraction of the hamstrings for 5 seconds. Three stretch-contraction cycles are completed. One researcher maintains the stretch position, while a second researcher controls the stretching and contraction times.
  Interventions: Other: Contract-Relax PNF (crPNF)
- Neuromuscular Electrical Stimulation (NMES + crPNF) (Experimental): The participants follow the same stretching protocol but with neuromuscular electrical stimulation (NMES) added. Electrical stimulation (50Hz, 300 µs pulse width) is applied using an Enraf Nonius TensMed S82 device. Two 5x9 cm electrodes are placed on the hamstrings, and participants adjust the current to a moderate-strong, but painless, contraction. One researcher maintains the stretch, while another adjusts the current intensity and controls the timing of the stretching and contraction.
  Interventions: Other: Neuromuscular electrical stimulation (NMES); Other: Contract-Relax PNF (crPNF)

INTERVENTIONS:
Other: Neuromuscular electrical stimulation (NMES) — Neuromuscular electrical stimulation (NMES) is applied during an isometric contraction. The NMES uses a symmetrical biphasic rectangular pulse (50Hz frequency and 300 µs phase width) delivered through an Enraf Nonius TensMed S82 electrostimulator. Two 5x9 cm electrodes are placed on the hamstrings, and participants adjust the current to a moderate-strong, yet painless, contraction level. During the intervention, one researcher maintains the stretch position while another researcher controls the current intensity and monitors the timing of both stretching and contractions.
  Arms: Neuromuscular Electrical Stimulation (NMES + crPNF)
Other: Contract-Relax PNF (crPNF) — The crPNF Group engages in an isolated contract-relax proprioceptive neuromuscular facilitation (crPNF) stretching protocol. Participants are positioned in a long sitting posture with maximum knee extension until they feel a moderate-strong stretch sensation, without pain. Each stretch lasts for 20 seconds, followed by a 5-second maximal voluntary isometric contraction of the hamstrings. Participants complete three cycles of stretch and contraction. One researcher maintains the stretch position while a second researcher controls the timing of the stretching and contractions.

SUMMARY:
Hamstring muscle injuries are common in basketball and result in long periods of inactivity. This study aims to compare two different stretching programs to assess their effects on hamstring flexibility and, secondarily, on jumping ability in young basketball players. One program uses a special stretching technique called proprioceptive neuromuscular facilitation (PNF), while the other uses the same stretching but adds electrical stimulation (NMES).

DETAILED DESCRIPTION:
Hamstring strains are increasingly common in sports, particularly in football and professional basketball, where they are the fourth most frequent injury. Stretching, especially when combined with techniques like proprioceptive neuromuscular facilitation (PNF), is a key method used to reduce the risk of these injuries. PNF, which involves alternating stretches with muscle contractions, is widely regarded for improving muscle flexibility. Recently, stretching combined with neuromuscular electrical stimulation (NMES) has also shown promise for increasing flexibility. A variant of PNF called contract-relax PNF (crPNF) has been proposed, where NMES is applied during the contraction phase to further enhance flexibility gains. However, there are no studies on the short-term effects of crPNF and crPNF + NMES in young male basketball players, a group known for higher degrees of hamstring shortening.

This study aims to compare the short-term effects of crPNF and crPNF + NMES on hamstring flexibility in young male basketball players and assess whether one technique is superior to the other. A secondary goal is to determine if either stretching protocol negatively impacts vertical jump ability, an important skill in basketball.

ELIGIBILITY:
Inclusion Criteria:

* Active basketball players who train at least 3 days a week
* Ages between 11 and 18 years
* Male gender

Exclusion Criteria:

* Participation in an organized hamstring stretching program
* Presence of low back pain
* Hamstring muscle injuries in the last 6 months
* Spinal or abdominal surgeries in the last 6 months

Ages: 11 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
The Popliteal Angle Test | Before and inmediately after the intervention
  The Popliteal Angle Test is validated for measuring hamstring extensibility. Participants are placed in the supine position. A researcher holds the hip at a 90° flexion and passively extends the knee until the participant feels a strong stretch without pain. The examiner records the knee extension degrees at that moment using an inclinometer. The test is repeated three times, and the average is obtained. A full knee extension corresponds to a value of 0 degrees, and a higher number of degrees indicates greater hamstring shortening.
The Sit & Reach Test | Before and inmediately after the intervention
  The Sit & Reach Test has high intra-examiner reliability and is validated for measuring hamstring extensibility. For its execution, participants are placed in a long sitting position with the soles of their feet against the base of the measurement box. Keeping their knees extended, they reach for the maximum possible distance in the box with their fingers. The test is repeated three times, and the average is obtained. Values are recorded in centimeters, where a greater distance indicates a higher degree of hamstring extensibility.

SECONDARY OUTCOMES:
The Counter Movement Jump | Before and inmediately after the intervention
  The Counter Movement Jump is validated and standardized in adolescents for measuring jumping ability. The instructions by Petrigna et al. are followed to perform the jump (Figure 2C). The My Jump App is used, which has high reliability and validity for measuring vertical jump height in centimeters. A greater height indicates a greater jumping ability.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Francisco Lisón Párraga, Dr, Principal Investigator — Cardenal Herrera University
Locations (1):
- University Ceu Cardenal Herrera, Alfara del Patriarca, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided